CLINICAL TRIAL: NCT03778112
Title: Prospective Evaluation of Multi-Parametric MRI Guided Stereotactic Body Radiotherapy (SBRT) for Localized Prostate Cancer
Brief Title: MRI Guided SBRT for Localized Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Dian Wang, Principal Investigator, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mpMRI SBRT Prostate | 15060207; 15060207 (Other: Rush University Medical Center)
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Results first posted 2023-02-14 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radiotherapy; SBRT; Stereotactic Body Radiotherapy; MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Negative mpMRI Prostate Scan (Experimental): SBRT to the whole prostate
  Interventions: Radiation: SBRT to whole prostate
- Positive mpMRI Prostate Scan (Experimental): IMRT to the prostate + seminal vesicles followed by SBRT boost to the whole prostate with SIB to MRI defined intraprostatic lesions
  Interventions: Radiation: IMRT followed by mpMRI guided SBRT boost with SIB to intraprostatic lesions

INTERVENTIONS:
Radiation: SBRT to whole prostate — Those patients with negative mpMRI prostate scan (PI-RADS 0-2) will receive SBRT (36.25 Gy/5 fractions) to the whole prostate
  Arms: Negative mpMRI Prostate Scan
Radiation: IMRT followed by mpMRI guided SBRT boost with SIB to intraprostatic lesions — Patients with positive or equivocal mpMRI prostate scan (PI-RADS 3-5) will receive IMRT (45 Gy/25 fractions) to the prostate + seminal vesicles +/- lymph nodes followed by SBRT boost (18 Gy/3 fractions) to the whole prostate with simultaneous integrated boost (21 Gy/3 fractions) to MRI defined intraprostatic lesions
  Arms: Positive mpMRI Prostate Scan

SUMMARY:
This study utilizes advanced imaging techniques (mpMRI prostate scan) to select and stratify patients for two different radiotherapy regimens based on the presence/absence of identifiable intraprostatic lesions.

In patients without identifiable prostate cancer lesions, SBRT to the prostate in 5 sessions (fractions) will be administered.

In patients with MRI-identified lesion(s), pelvic IMRT in 25 fractions will be administered followed by an SBRT prostate boost while simultaneously treating the prostate cancer lesion(s) to a higher dose in 3 fractions.

DETAILED DESCRIPTION:
Radiotherapy (RT) is considered standard of care treatment for prostate cancer. Conventional RT regimens consist of 8-9 weeks of daily RT. Recent data support the use of hypofractionated RT (5-6 weeks) due to similar disease control in a contracted treatment time. This study combines the benefits of RT dose escalation while shortening the overall RT treatment course.

In this protocol, patients will undergo a pretreatment mpMRI prostate scan and be stratified to two separate SBRT regimens depending on whether prostate lesions are present. For patients without any positive mpMRI lesions, an SBRT monotherapy (36.25 Gy in 5 fractions) approach will be utilized. Patients with an equivocal or positive mpMRI lesion(s), will receive IG-IMRT (45 Gy in 25 fractions) to prostate and seminal vesicle +/- lymph nodes followed by a SBRT whole prostate boost (18 Gy in 3 fractions) with a simultaneously integrated boost (SIB) (21 Gy in 3 fractions) to intraprostatic lesion(s) only.

Patients will be regularly assessed every 3 months for the first 2 years and then every 6 months, indefinitely. Side effects will be monitored using the standardized international prostate symptom score (I-PSS) and Sexual Health Inventory of Men (SHIM) questionnaires at baseline and subsequent follow-up appointments.

Hypothesis: MRI-guided treatment planning and delivery can selectively target high-risk prostate cancer nodules and deliver a higher effective RT dose, to achieve maximal tumor control without increasing toxicity, all in a shortened treatment duration.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate adenocarcinoma within 1 year of randomization
* NCCN Low to High Risk localized prostate cancer
* Zubrod Performance Status 0-1 within 60 days prior to registration

Exclusion Criteria:

* Prior or concurrent invasive malignancy (except non-melanoma skin cancer)
* Regional Lymph Node (N1) involvement
* Distant Metastases (M1) involvement
* History of prior pelvic irradiation (external beam radiotherapy or brachytherapy)
* Prior chemotherapy
* Severe, active co-morbidities (unstable angina and/or CHF; MI; COPD; liver disease; AIDS)
* Acute bacterial or fungal infection requiring IV antibiotics
* Inability to undergo MRI
* Inability to receive fiducial markers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2029-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dian Wang, MD, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Negative mpMRI Prostate Scan | Positive mpMRI Prostate Scan
Started | 4 | 50
Completed | 4 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative mpMRI Prostate Scan | Positive mpMRI Prostate Scan | Total
Number analyzed (Participants) | 4 | 50 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 16 | 18
  >=65 years | 2 | 34 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 50 | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 50 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Late Radiation Induced Genitourinary and Gastrointestinal Toxicity
Description: Number of Participants with late grade 3-5 genitourinary and gastrointestinal toxicity following mpMRI guided radiation treatment. Late toxicity will be defined as toxicity occurring more than nine months from the start of radiotherapy.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Negative mpMRI Prostate Scan | Positive mpMRI Prostate Scan
Number analyzed (Participants) | 4 | 50
participants | 4 | 50

2. Secondary Outcome: Number of Participants With Acute Radiation Induced Genitourinary Adverse Event
Description: Adverse acute events are evaluated by the CTEP Active Version of the NCI CTCAE. The treatment-related attribution includes definitely, probably or possibly related to treatment. An acute adverse event is defined as the first occurrence of worst severity of the adverse event ≤30 days after the completion of RT. For each cohort, we will evaluate the acute radiation therapy-related adverse events. Specifically, we are interested in the percentage of acute GI and GU Grade 3+ adverse events that occur in each arm, which is considered to be similar to the high RT dose arm of RTOG 0126 in terms of RT dose. For this arm, a reported 1% of patients experienced Grade 3+ GI/GU acute toxicity, with no patient experiencing Grade 4 or 5 toxicities. If either hypofractionated arm has an acceptable percentage, then that arm will be deemed to have an acceptable adverse event profile. We will report the percentage for each arm as well as the one-sided 97.5% confidence interval.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Negative mpMRI Prostate Scan | Positive mpMRI Prostate Scan
Number analyzed (Participants) | 4 | 50
participants | 4 | 50

3. Secondary Outcome: Biochemical Recurrence
Description: Biochemical (PSA) recurrence is defined according to the proposed new Radiation Therapy Oncology Group/American Society for Therapeutic Radiology and Oncology (RTOG-ASTRO) criteria also known as the RTOG Phoenix definition: an increase of the PSA level at least 2 ng/mL greater than the minimum level reached after therapy (lowest PSA+ 2 criterion). PSA failure at 1, 2, and 5 years will be estimated for each cohort by the cumulative incidence method.
Time Frame: 18 months
Reporting Status: Not Posted

4. Secondary Outcome: Disease Free-Survival
Description: The disease-free survival duration will be measured from the date of registration to the date of documentation of disease progression or until the date of death from any cause. DFS at 1, 2, and 5 years will be estimated for each c o h o r t by the Kaplan-Meier method. Also, 95% confidence intervals will be reported.
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data collected up to 54 months from registration.
Arm/Group | Negative mpMRI Prostate Scan | Positive mpMRI Prostate Scan
All-Cause Mortality (participants affected / at risk) | 0/4 | 4/50
Serious Adverse Events (participants affected / at risk) | 4/4 | 50/50
Other Adverse Events (participants affected / at risk) | 0/4 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Negative mpMRI Prostate Scan (N=4) | Positive mpMRI Prostate Scan (N=50)
Other acute/late grade 1-2 GI/GU event (Gastrointestinal disorders) | 4 (4) | 48 (48)
grade late GU toxicity (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT03778112/Prot_SAP_001.pdf
  • Informed Consent Form (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT03778112/ICF_000.pdf